CLINICAL TRIAL: NCT07323134
Title: The Effect of Semaglutide on the Intestinal Flora in Obesity
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-science-480
Record Dates: First submitted 2025-07-13; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Semaglutide Injection — Semaglutide Injection

SUMMARY:
For obese individuals, semaglutide treatment was adopted. By using multi-omics techniques such as fecal metagenomic sequencing and based on in vitro strain screening platforms, the effects and specific mechanisms of semaglutide on the intestinal flora of obese patients were clarified.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old;
* BMI ≥ 30kg/m²;
* At least one self-reported history of unsuccessful lifestyle weight loss;
* Subjects who agree to participate in the project and sign the informed consent form.

Exclusion Criteria:

* Weight changes within 3 months prior to screening (self-reported) >5%;
* Having received any drug treatment for obesity within the three months prior to screening;
* The application of hypoglycemic drugs within 3 months before screening, or HbA1c≥ 6.5%, or a history of type 1 or type 2 diabetes;
* Participants who have received treatment with immunosuppressants, steroids, antidiarrheal drugs, antibiotics, probiotics, lipid-lowering drugs and/or other gastrointestinal motility drugs within 3 months prior to screening;
* Previously diagnosed overweight or obesity due to endocrine causes, such as Cushing's syndrome, etc;
* Triglycerides ≥500mg/dL (5.65mmol/L) during screening;
* It is known that there are clinically significant gastric emptying abnormalities (e.g., severe diabetic gastroparesis or gastric outlet obstruction), a history of gastrointestinal diseases and surgical history;
* Abnormal thyroid function;
* History of mental illness;
* History of multiple endocrine tumors or medullary thyroid cancer, family history, or calcitonin ≥6pg/mL;
* Abnormal liver function during screening, that is, alanine aminotransferase and/or aspartate aminotransferase > 3*ULN;
* Abnormal renal function during screening, that is, the estimated glomerular filtration rate is less than 60mL/min/1.75m2;
* History of cardiovascular diseases;
* History of malignant tumors;
* Pregnancy or lactation;
* As determined by the researcher, there are other physical, psychological or other conditions that make one unsuitable to participate in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese patients who visited the Department of Endocrinology of Beijing Chaoyang Hospital Affiliated to Capital Medical University
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The composition of the gut microbiota changes relative to the baseline | Baseline,4weeks,8weeks,12weeks
  The changes in the composition of the gut microbiota in obese individuals after 12 weeks of semaglutide treatment relative to the baseline (baseline is defined as the composition of the gut microbiota at the time of enrollment), including alterations in gut microbiota abundance and Shannon diversity index (α -diversity), etc.

DOCUMENTS (1):
  • Study Protocol (2025-04-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT07323134/Prot_000.pdf